CLINICAL TRIAL: NCT03371160
Title: A Feasibility Study to Evaluate the Clinical Safety of Nutriseal™ Enteral Feeding Tube Placement Using the Nutriseal™ Nutriplace™ System in Patients
Brief Title: Feasibility Study to Evaluate Safety of Nutriseal™ Nutriplace™ System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Nutriseal L.P (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NUTRI001
Record Dates: First submitted 2017-12-01; First posted 2017-12-13 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Nutriplace™ System (Experimental): Placement of the Nutriseal™ Enteral Feeding Tube in the stomach or small intestine of adult patients who require feedings via the oro/nasoenteric route, using the Nutriplace™ System.
  Interventions: Device: Nutriplace™ System

INTERVENTIONS:
Device: Nutriplace™ System — The Nutriseal™ Nutriplace™ System is an electromagnetic tracking system for feeding tube placement designed to aid qualified operators in the placement of the Nutriseal™ Enteral Feeding Tube™ into the stomach or small intestine.

SUMMARY:
This is a single center, non-randomized feasibility clinical evaluation that is designed to affirm the safety of the Nutriplace™ System guidance during the placement of the Nutriseal™ enteral feeding tubes.

DETAILED DESCRIPTION:
Enteral nutrition is the preferred route for the provision of nutritional support in most critical ill patients with functional gastrointestinal tract. Achieving early enteral nutrition (EN) in critically ill patients is associated with fewer major complications, reduced mortality and length of hospital stay, and significant cost savings.

It is estimated that approximately 1.2 million feeding tubes are placed blindly each year in the United States alone. Despite the obvious advantages of the enteral tube feeding, inadvertent placement of enteral feeding tube (EFT) into the airway is relatively common and can result in significant pulmonary injury including pneumothorax and pneumonia. Airway misplacement occurs in 1.2-4 % of blind EFT insertions, with 0.2 to 1.2% of all the feeding tube placements cause pulmonary complications to patients.

The gold standard for detecting inadvertent placement of a feeding tube in the lungs is radiography. However, because of its cost, possible delay of feedings while waiting for radiography, and risk for radiation exposure, clinicians continue to seek for alternative methods to confirm correct placement.

All the above mentioned, emphasizes the fact that safe and effective delivery of nasoenteral tube feedings requires assurance that the feeding tube tip is in a proper position.

The Nutriplace™ System is an electromagnetic tracking system which tracks the path of the feeding tube during placement.

The benefit of the system when EFT is misdirected into the pulmonary system is a real-time visual tracing, which may prompt users to withdraw the tube and reinsert it.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be >21 years of age
2. Patients must require placement of a nasoenteral feeding tube
3. Patients have an endotracheal tube, OR Do not have an endotracheal tube but are sedated (RASS score of -2 or less) and/or obtunded (Glasgow Coma scale of 9-12)
4. Patients or legal authorized representative must be able to understand and adhere to all protocol procedures and be willing and able to provide written informed consent

Exclusion Criteria:

1. Patients must not have a history of:

   * Esophageal varices or ulcers
   * Upper airway obstruction
   * Upper GI stenosis or obstruction
   * Trauma involving sinuses, nares face or neck that would prevent Nasogastriv (NG) tube insertion
   * Deformities of the sinus cavities and/or skull base
   * Esophageal cancer or neoplasm
2. Patients must not have a significant concomitant illness that would adversely affect their participation in the study
3. Female patients who are pregnant or lactating

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: May Olayan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nutriplace™ System: Placement of the Nutriseal™ Enteral Feeding Tube in the stomach or small intestine of adult patients who require feedings via the oro/nasoenteric route, using the Nutriplace™ System.
  Nutriplace™ System: The Nutriseal™ Nutriplace™ System is designed to aid qualified operators in the placement of the Nutriseal™ Enteral Feeding Tube™ into the stomach or small intestine.
Period: Overall Study
Arm/Group | Nutriplace™ System
Started | 22
Completed Data Collection of Primary Endpoint | 14
Completed | 14 (Of 22 enrolled participants, 19 met inclusion/ exclusion criteria and underwent a tube placement attempt. From these 22 participants, 14 completed a successful tube placement.)
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Nutriplace™ System
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 62.5 [23 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 5
  White | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successfully Placed Enteral Feeding Tube
Description: Enteral tube (EFT) can be placed in the correct anatomical position without occurrence of guidance-related adverse events.
  Procedure success was evaluated by comparing tube tip location according to the NUTRIPLACE System and abdominal and/or thoracic X-Ray.
  Guidance-related AEs were evaluated through the documentation of any guidance-related serious adverse events (SAE) or adverse events (AE) occurring during a subject's participation in the study.
Time Frame: During procedure visit
Population: Of 22 enrolled participants, 19 met inclusion/ exclusion criteria and underwent a tube placement attempt. From these 22 participants, 14 completed a successful tube placement using the ENvue system.
  The study was halted pre-maturely due to a very low enrollment rate at the site.
Measure: Count of Participants; unit: Participants
Arm/Group | Nutriplace™ System
Number analyzed (Participants) | 22
Participants | 14

2. Secondary Outcome: Number of Participants Requiring Replacement and/or Repositioning of the Feeding Tube
Description: Number of placement attempts was evaluated by number of replacement and repositioning events, as defined below:
  * Replacement: Complete removal of the tube from the patient or retraction above the level of the pharynx followed by reinsertion
  * Repositioning: Changing position of tube without complete removal of the tube
Time Frame: During procedure visit
Measure: Count of Participants; unit: Participants
Arm/Group | Nutriplace™ System
Number analyzed (Participants) | 14
Participants | 10

3. Secondary Outcome: Number of Participants Reporting Retrograde Tube Migration in the Follow-up Visit
Description: Tube Migration was defined as: Retrograde migration from desired placement position
Time Frame: During follow-up visit (20-48 hours post tube placement
Measure: Count of Participants; unit: Participants
Arm/Group | Nutriplace™ System
Number analyzed (Participants) | 12
Participants | 1

ADVERSE EVENTS:
Time Frame: From the participant's tube placement procedure (day 0) to the end of of the follow-up visit (20-48 hours post tube placement)
Description: Analysis was performed on all subjects that underwent a tube placement attempt (19 subjects)
Arm/Group | Nutriplace™ System
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed. Twelve months following the completion of the study, Investigator may publish the results of the study. Investigator shall provide sponsor advanced copies of any proposed publication sixty days prior to planned publication Sponsor will have sixty days to review the proposed publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03371160/Prot_SAP_000.pdf